CLINICAL TRIAL: NCT04765436
Title: A Phase I, First-in-Human, Observer-Blinded, Randomized, Placebo Controlled, Ascending Dose Study to Evaluate the Safety, Tolerability, and Immunogenicity of PTX-COVID19-B Vaccine in Healthy Seronegative Adults Aged 18-64
Brief Title: PTX-COVID19-B, an mRNA Humoral Vaccine, is Intended for Prevention of COVID-19 in a General Population. This Study is Designed to Evaluate Safety, Tolerability, and Immunogenicity of PTX-COVID19-B Vaccine in Healthy Seronegative Adults Aged 18-64
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Therapeutics Holdings Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-CL-001
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Covid19 Vaccine
MeSH Terms: interventions — PTX-COVID19-B COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTX-COVID19-B (Experimental): Participants, 45 healthy adults 18 to 64 years of age, will receive 1 intramuscular (IM) injection of PTX-COVID19-B vaccine in doses of 16 μg, 40 μg and 100 μg on Day 1, followed by a second dose on Day 28, respectively.
  Interventions: Biological: PTX-COVID19-B
- Placebo (Placebo Comparator): Participants, 15 healthy adults 18 to 64 years of age, will receive 1 IM injection of matching placebo on Day 1, followed by a second dose on Day 28.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PTX-COVID19-B — Sterile solution for injection
  Arms: PTX-COVID19-B
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The Vaccine Product, PTX-COVID19-B mRNA Humoral Vaccine, is intended for prevention of COVID-19 in a general population. This study is designed to evaluate the safety, tolerability, and immunogenicity of PTX-COVID19-B vaccine in healthy seronegative adults aged 18 to 64.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all inclusion criteria to be eligible for study participation. In addition, racial and ethnic minorities will be sought to obtain a diverse study population.

1. Subject has read, understood, and signed the informed consent form.
2. Healthy adult males and females 18 to 64 years of age, inclusive, at screening
3. Seronegative to SARS-CoV-2 and reverse transcription-polymerase chain reaction (RT-PCR)-negative at screening, without evidence of recent of exposure or viral respiratory disease not identified as influenza or RSV (febrile or lower respiratory tract infection)
4. Body mass index of ≥ 18 and ≤ 30 kg/m2 at screening
5. Must be in general good health before study participation with no clinically relevant abnormalities that could interfere with study assessments.
6. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception (i.e., including hysterectomy, bilateral salpingectomy, and bilateral oophorectomy, hormonal oral [in combination with male condoms with spermicide], transdermal, implant, or injection, barrier [i.e., condom, diaphragm with spermicide]; intrauterine device; vasectomized partner [6 months minimum], clinically sterile partner; or abstinence) during the study.

   * A female subject is considered a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile.
   * Subjects not of childbearing potential are not required to use any other forms of contraception during the study. Non-childbearing potential is defined as subject confirmed:

     * Surgical sterilization (e.g., bilateral oophorectomy, bilateral salpingectomy, bilateral occlusion by cautery [Essure System® is not acceptable], hysterectomy, or tubal ligation)
     * Postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to screening); if postmenopausal status is unclear, pregnancy tests will be performed prior to vaccinations.
7. Women of childbearing potential must have a negative pregnancy test before each vaccination. If menopausal status is unclear, a pregnancy test is required.
8. Must be able to attend all visits (scheduled and unscheduled, as applicable) for the duration of the study and comply with all study procedures, including daily completion of the Diary Card after each injection.

Exclusion Criteria:

Subjects will not be eligible for study participation if they meet any of the exclusion criteria, or will be discontinued at the discretion of the investigator if they develop any of the exclusion criteria during the study.

1. History of an acute or chronic medical condition including dementia that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses.
2. History of any medical conditions that place subjects at higher risk for severe illness due to SARS-CoV-2 will be excluded including:

   * Chronic kidney disease
   * COPD (chronic obstructive pulmonary disease)
   * Heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
   * Any Immunocompromised state including from transplantation, history immunodeficiency, HIV, immunosuppressive drug intake.
   * Sickle cell disease
   * Current smoker or history of >5 pack/years of smoking.
   * Type 2 diabetes mellitus

   Subjects with history of any of the following conditions might be at an increased risk of complications from Covid 19 and will be excluded:
   * Asthma (moderate-to-severe)
   * Cerebrovascular disease (affects blood vessels and blood supply to the brain)
   * Cystic fibrosis
   * Hypertension or high blood pressure
   * Neurologic conditions, such as dementia
   * Liver disease
   * Pulmonary fibrosis (having damaged or scarred lung tissues)
   * Thalassemia (a type of blood disorder)
   * Type 1 diabetes mellitus
3. History of ongoing clinical condition or medication or treatments that may adversely affect the immune system.
4. Individuals who are seropositive or RT-PCR positive for SARS-CoV-2, including prior to a second dose of PTX-COVID19-B vaccine.
5. Individuals who are at increased risk of exposure to SARS-CoV-2 (e.g., healthcare workers, emergency responders).
6. Close contact of anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration.
7. Living in a group setting or group care facility (e.g., dormitory, assisted living or nursing home).
8. Individuals with any elevated (Grade 1 or higher) laboratory test assessed as clinically significant for age/sex by the investigator at screening.
9. Individuals with any elevated for age/sex (Grade 1 or higher) liver function enzyme at screening, regardless of the appraisal of clinical significance (one retest permitted). The criteria for excluding subjects with elevated liver enzymes are as follows:

   * Alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, or gamma-glutamyl transferase > 1.5 × upper limit of normal (ULN)
   * Total bilirubin > 1.5 × ULN
10. Active neoplastic disease (excluding nonmelanoma skin cancer that was successfully treated) or a history of any hematological malignancy. "Active" is defined as having received treatment within the past 5 years.
11. Long-term (> 2 weeks) use of oral or parenteral steroids or high-dose inhaled steroids (> 800 μg/day of beclomethasone dipropionate or equivalent) within 6 months before screening (nasal and topical steroids are allowed).
12. History of autoimmune, inflammatory disease, or PIMMCs.
13. Women currently pregnant, lactating, or planning a pregnancy between enrollment and 181 days after randomization.
14. History of Guillain-Barré Syndrome or any degenerative neurology disorder.
15. History of anaphylactic-type reaction to any injected vaccines.
16. Known or suspected hypersensitivity to 1 or more of the components of the vaccine.
17. History of alcohol abuse, illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of screening.
18. Acute illness or fever (temperature >37.5C) within 3 days before study enrollment (enrollment may be delayed for full recovery if acceptable to the investigator).
19. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month (3 months for immunoglobulins) before enrollment in this study; or who expect to receive another experimental agent during participation in this study.
20. Receipt of immunoglobulin or another blood product within the 3 months before enrollment in this study or those who expect to receive immunoglobulin or another blood product during this study.
21. Individuals who intend to donate blood within 6 months after the first vaccination and within 30 days post the last donation from Visit 1.
22. Individuals using prescription medications for prophylaxis of SARS-CoV-2.
23. Individuals who plan to receive another vaccine within the first 3 months of the study except influenza vaccine which should not be given within 2 weeks of vaccine.
24. Receipt of any other SARS-CoV-2 or other experimental coronavirus (Middle East Respiratory Syndrome, SARS etc.) vaccine at any time prior to or during the study.
25. Receipt of any investigational vaccine or investigational drug within 1 month of enrollment and through the end of the study (1 year after the last vaccination).
26. Plan to travel outside Canada from enrollment through Day 42.
27. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
28. Significant blood loss (> 400 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
29. Strenuous activity or significant alcohol intake (as assessed by the investigator) within 72 hours prior to safety laboratory sample collection.
30. Positive urine drugs of abuse screen.
31. Positive screen for human immunodeficiency virus-1 and -2 antibodies, hepatitis B surface antigen, or hepatitis C virus antibody.
32. Involved in the planning or conduct of this study.
33. Unwilling or unlikely to comply with the requirements of the study.
34. Subjects is an employee, contractor, or friend or relative of any employee of sponsor, CRO, study site, or site affiliate.
35. Subjects oximetry is <90%

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) during the follow-up after each vaccination | Day 1 through Day 3
  Daily solicited adverse events will be analyzed using both the Per Protocol (PP) and Safety Populations.
Assessments of AEs | Day 1 through Day 42
  Reports of unsolicited AEs
Assessment of Safety | Day 1 through Day 395
  Reports of Medically attended AEs
  Reports of serious adverse events (SAEs)
  Reports of adverse events of special interest
  Reports of potential immunemediated medical conditions
Immunogenicity analysis | Day 1 and Day 28
  Cell-mediated immunity using blood/peripheral blood mononuclear cells (PBMCs [Flow Cytometry Assay])
  Antibodies (anti-COVID-19 immunoglobulin (Ig), IgG, IgA [enzyme-linked immunosorbent assay]; and anti-COVID-19 neutralization titer assays)

CONTACTS AND LOCATIONS:
Locations (1):
- Manna Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Orozco N, Vale N, Mihic A, Amor T, Reiter L, Arita Y, Samson R, Hu Q, Gingras AC, Sorenson BT, Marcusson EG, Patel P. Phase I randomized, observer-blinded, placebo-controlled study of a SARS-CoV-2 mRNA vaccine PTX-COVID19-B. Sci Rep. 2023 May 26;13(1):8557. doi: 10.1038/s41598-023-35662-y. PMID 37236995